CLINICAL TRIAL: NCT04581083
Title: Validation of Laboratory Techniques, Strategies, and Types of Samples for Epidemiological Control in the Covid-19 Pandemic, Tarija-Bolivia
Brief Title: Validation of Laboratory Techniques, Strategies, and Types of Samples for Epidemiological Control in the Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Hunter College of City University of New York (Other)
Collaborators: Universidad Autonoma Juan Misael Saracho (Unknown); Gobierno Autonomo Departamental De Tarija (Unknown); SEDES - Tarija (Unknown); CAINCO - Bolivia (Unknown); Universidad Mayor de San Simon (Unknown)
Responsible Party: Principal Investigator, Rodrigo Arce Cardozo, Adjunct Assistant Professor, Hunter College of The City University of New York
Other Study IDs: PROY - UAJMS001/2020
Record Dates: First submitted 2020-10-07; First posted 2020-10-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Covid19
Keywords: COVID 19; Bolivia; Clinical Laboratory Techniques
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — nasopharyngeal swab and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volunteer participants: Samples of volunteer participants will be collected after informed consent and classified as symptomatic, asymptomatic and negative.
  Interventions: Diagnostic Test: RT-PCR; Diagnostic Test: LAMP; Diagnostic Test: POOL RT-PCR; Diagnostic Test: POOL LAMP

INTERVENTIONS:
Diagnostic Test: RT-PCR — RT-PCR (Gold standard): Real-time PCR testing with reverse transcriptase (RT-PCR). The test consists of a polymerase chain reaction that has previously had a reverse transcription phase, RT. This test allows the cADN (complementary DNA) to be obtained from a RNA chain. This technique allows the detection and amplification of a sequence from a strand of RNA.
  Other Names: Real-Time Polymerase Chain Reaction
Diagnostic Test: LAMP — LAMP: The LAMP technique, like PCR, has the ability to amplify specific DNA fragments (target sequence), allowing for highly sensitive detection of pathogens. Unlike pcr, LAMP requires between 4 and 6 feeders, external F3 and B3 feeders, which hybridte with the outer regions of the target sequence, while the internal FIP and BIP have sequences in both ways that allow the formation of a loop. The LAMP reaction is isothermal, i.e. it takes place at a single temperature. LAMP has been successfully used to detect viral diseases as well as viral pathogens such as West Nile virus, TMR-1, Norovirus, avian influenza, foot-and-mouth disease, classical swine fever, among others.
  Other Names: Loop-mediated isothermal amplification
Diagnostic Test: POOL RT-PCR — POOL RT-PCR: This test aims to mix in a single sample the extractions obtained from several people. The joint sample is evaluated and, if negative, it is understood that all are free of COVID-19; if it is positive, an array system is used to detect the affected person. That is, a single PCR (polymerase chain reaction), the diagnostic test used to detect the virus pathogen is applied to a group and repeated individually if positive.
  Other Names: Pooled Real-Time Polymerase Chain Reaction
Diagnostic Test: POOL LAMP — POOL LAMP: Like the RT-PCR pool test. This test essentially involves mixing in a single sample the extractions obtained from several people. This joint sample is tested and, if it is negative, it is understood that everyone is free of COVID-19; if it is positive, an array system is used to detect the affected person. That is: a single LAMP applies to a group
  Other Names: Pooled Loop-mediated isothermal amplification

SUMMARY:
This is a study of validation for diagnostic techniques used on epidemiological control in the COVID-19 pandemic. It will be carried out in accredited public, private and university clinical laboratories of the collaborator institutions of the project based in Tarija, Bolivia. It is designed as a sectional validation study, using samples from specific groups of participants from the municipality of Tarija grouped according to their category with respect to symptoms and viral load of COVID-19. The sample is selected for convenience.

ELIGIBILITY:
Inclusion criteria:

* Symptomatic: Subjects with signs and symptoms of respiratory infection less than or equal to 3 days, preferably with clinical and molecular diagnosis compatible with Covid-19.
* Asymptomatics: Subjects who have had direct contact with people infected and who have not shown any symptoms related to Covid-19.
* Negative: Individuals with negative RT-PCR testing for SARS-CoV-2 (reference test) who have not manifested any symptoms seven days prior to sampling.

Exclusion criteria:

* Adults under the age of 21 or over 65
* Subjects with a clinical history of autoimmune disease or chemotherapy treatments.
* Subjects who have received transfusions or convalescent plasma in the last month prior to enrollment.
* Subjects with prior diagnosis of other infectious diseases such as, but not limited to AIDS, Hepatitis B or C, Tuberculosis, or any other ongoing or unresolved diseases.
* Subjects with malformation or oncological pathology of the upper respiratory track that may hinder sample collection, including but not limited to deviated septum, allergic rhinitis.
* Subjects who have not signed or can not sign the informed consent form
* Subjects not able to provide their complete information or access to their clinical history.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Validation will be carried out using samples from volunteer adults from the municipality of Tarija, Bolivia, without gender restriction. Samples will be grouped according to the clinical classification determined above. These individuals will need to sign the informed consent form required to agree to be part of the study and provide their complete information or access to their medical history.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Validation | 1 month
  Validate different molecular tests and sampling and sample type strategies used in epidemiological control of COVID-19 diagnosis in Tarija, Bolivia.

SECONDARY OUTCOMES:
RT- PCR (Saliva) | 1 week
  Validate the use of molecular testing based on the PCR method using Saliva samples
LAMP | 1 week
  Validate the use of the molecular test based on the LAMP method using saliva and nasopharyngeal samples
POOL PCR | 1 week
  Validate the use of molecular tests with Pool PCR strategy using saliva samples
POOL LAMP | 1 week
  Validate the use of molecular tests with Pool LAMP strategy using saliva samples

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Shoji, PhD, Principal Investigator — Galapagos NV; Rodrigo Arce Cardozo, MD, MPH, Study Chair — City University of New York, School of Public Health
Locations (1):
- Universidad Autónoma Juan Misael Saracho, Tarija, Bolivia

IPD SHARING:
Plan to Share IPD: Yes
We will share deidentified data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Paper submitted for publication
Access Criteria: Open

REFERENCES:
- See also: Local Sponsor University Website — https://www.uajms.edu.bo/